CLINICAL TRIAL: NCT03518710
Title: Vision, Attention and Reading in Neurofibromatosis Type 1 (NF1) Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/17/0376; 2017-A02907-46 (Other: UHToulouse)
Record Dates: First submitted 2018-04-23; First posted 2018-05-08 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Neurofibromatosis Type 1
Keywords: child; reading; vision; attention; therapeutical perspectives
MeSH Terms: conditions — Neurofibromatosis 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with NF1 (Experimental): One experimental group of NF1 children with 3 reading levels (1st grade, 2nd grade and 3rd grade). For this research they will pass :
  * Neuropsychological evaluation
  * Evaluation of the reading assistance technique
  Interventions: Other: Neuropsychological evaluation; Other: Evaluation of the reading assistance technique

INTERVENTIONS:
Other: Neuropsychological evaluation — Neuropsychological evaluation (about 60 min) the same day realized by a student in Science Thesis under the responsibility of Prof. Yves Chaix and including:
  * Process evaluation:
  * Oculomotors: DEM test (5min)
  * Visuo-attention: computerized STROOP (15min)
  * Visuo-Perceptive: DTVP3 (30min)
  * Phonological & lexical: Exalang (10min)
Other: Evaluation of the reading assistance technique — Evaluation of the reading assistance technique (about 30 min) and comprising:
  - Reading evaluation:Test lark (3min) Experimental task: 3-way help with reading (without help, color help and highlight help (25 min)

SUMMARY:
The present project will therefore focus upon those processes related to visual attention and perceptual abilities and on their potential to explain reading behavior and reading problems in NF1. The main objective of this study is to clarify the specificity and heterogeneity of reading profiles and the causes of its disturbance in NF1. In particular, this project allow the investigators to study more precisely the relations between perceptual, oculomotor and visuo-attentional skills in NF1 children and reading abilities. In addition, a new oculomotor/perceptual reading aid for NF1 children will be evaluated. The investigators believe that the early intervention for perceptual, visuo-attentional or oculomotor problems may promote academic skill development.

DETAILED DESCRIPTION:
Although some NF1 children manage in the end to exhibit "expert" reading behavior, a non-negligible number of them have real problems learning this skill. Today's estimates indicate that 30-60% of NF1 children suffer from written-language learning disorder. Studies of the effects of the neurocognitive deficit on academic performance are relatively rare, owing to the small size of the populations concerned. However, research is needed to develop effective rehabilitation programs. At the current time, most tools available to professionals are designed for the evaluation and remediation of child language problems, particularly difficulties related to the acquisition of meta-phonological skills. The findings from dyslexics and typically developing readers however suggest a strong relationship between reading ability and visual processing. The main goal of this study is to investigate the occurrence of perceptual, visuo-attentional and oculomotor deficits in NF1 children and their potential to explain reading behavior and reading problems in this population. The investigators hope to contribute to the process of clarifying the specificity and heterogeneity of reading profiles and the causes of its disturbance in NF1. The second objective of the study is to evaluate an oculomotor/perceptual reading aid for NF1 children; in particular, the idea of the training is to help the readers to land their saccades at the optimal viewing position1 (OVP) of each word (highlighting the letter at the OVP or putting it in color, so that the saccades they make would land near the centre of the word, at the OVP). Eye movement control during reading is a highly automated process; people are not aware of most of the saccades and fixations they make. This tool is a way to train children to control these subconscious saccades and fixations. Note that, our team has already demonstrated the usefulness of this reading aid for beginning readers. This project have important implications from a clinical perspective, by providing the opportunity to gain insight into the reading difficulties of NF1 children, in view of establishing thorough and accurate assessment procedures and proposing child-specific guidelines and remediation methods that take into account the particular processes affected. Providing a clearer picture of visuo-attentional and perceptual skills in children with NF1 would be of considerable clinical benefit, not least for supporting targeted clinical practices. Moreover, NF1 children could benefit from a new remediation tool that allow them to have feedback on their reading ability, and to read more easily, more rapidly, and with better comprehension. If appropriate interventions are implemented at an early age, academic skill development could be altered, preventing subtle learning difficulties from becoming more pronounced over time.

ELIGIBILITY:
Inclusion Criteria:

* Child with a NF1 following the clinically-based criteria agreed at the international Consensus Conference
* Age between 7 and 9 years old child in 1st - 3rd grades with 5 children/grade
* Informed children and written consent obtained from one of the parents or other lawful representative
* Child who is covered by the social security scheme

Exclusion Criteria:

* left-handed children
* associated neurological disorder such as brain tumors or epilepsy
* mental retardation (IQ <70 or Wechsler Intelligence Scale for Children (WISC) scores SIM et IC < 7)
* children with Autism Spectrum Disorder
* diagnosis of attention deficit hyperactivity disorder (ADHD) (DSM-IV), with presence of hyperactive-impulsive or inattentive symptom
* pharmaceutical treatment (e.g., anti-depressants, anxiolytics)

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the score obtained for Oculomotor Processes | 1 day
  The visual process : Oculomotor Processes : Vertical,Horizontal Time with the Ratio with the Developmental Eye Movement Test (DEM test) : a standard of evaluation oculomotor in children with reading difficulties
Evaluation of the composite score obtained for Visuo-perceptual process | 1 day
  The visual process : Visuo-perceptual process : it's a composite score : Composite score of perceptual treatment with pure visual perception score and visuo-motor integration with a Developmental Test of Visual Perception, 3rd (DTVP3) test is Visual perception development test
Evaluation of the score obtained : Visual-attentional process | 1 day
  Visual-attentional process : reaction time (milli Sec) with the percentage of correct answers to the computerized Stroop to show that attention is a selective process and that it is very difficult to read and name colors at the same time

SECONDARY OUTCOMES:
Alouette Reading Test | 1 day
  To evaluate language skills like phonological awareness with lexical stock Alouette Reading Test's aim is for the accuracy index and CTL speed index :The Alouette test is a reading test that evaluates the level of lexical decoding (automaticity). It consists of reading a standard text aloud and count the number of words read and errors in a given time

CONTACTS AND LOCATIONS:
Overall Officials: Yves Chaix, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No